CLINICAL TRIAL: NCT07276386
Title: Phase 2 Sequential Treatment With Melphalan/HDS Via Percutaneous Hepatic Perfusion Followed by Tebentafusp in the Treatment of Metastatic Uveal Melanoma
Brief Title: Phase 2 Combination of Melphalan/HDS Via PHP + Tebentafusp in Treating Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23724
Record Dates: First submitted 2025-12-01; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential PHP with Melphalan/HDS followed by Tebentafusp (Experimental): Patients will undergo two percutaneous hepatic perfusion (PHP) procedures with melphalan/HDS, spaced 6-8 weeks apart. Tebentafusp will be initiated within 6 weeks (+/- 2 weeks) after the second PHP and administered weekly for 1 year. Additional PHP procedures (up to 6 total) may be performed as standard of care if disease progression occurs while on tebentafusp.
  Interventions: Drug: Melphalan/HDS (Percutaneous Hepatic Perfusion); Drug: Tebentafusp

INTERVENTIONS:
Drug: Melphalan/HDS (Percutaneous Hepatic Perfusion) — 3 mg/kg ideal body weight (max 220 mg) infused via hepatic artery catheter.
Drug: Tebentafusp — 20 mcg IV day 1, 30 mcg day 8, 68 mcg day 15, then weekly thereafter.

SUMMARY:
This Phase 2 study evaluates the efficacy and safety of sequential treatment with percutaneous hepatic perfusion (PHP) using melphalan/HDS followed by tebentafusp in patients with metastatic uveal melanoma (mUM) with isolated liver metastases. The rationale is that PHP enhances antigen release and immunomodulation, potentially sensitizing tumors to tebentafusp in HLA-A*02:01-positive patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥18 years of age on the day of signing informed consent.
* ECOG performance status of 0 or 1.
* Histologically or cytologically confirmed liver metastasis of uveal melanoma.
* HLA-A*02:01 positive status.
* Measurable disease by computed tomography (CT) per RECIST 1.1 with at least one target lesion identified in the liver.
* Patient deemed suitable for PHP and tebentafusp.
* Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female patients of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male patients of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 150 days after the last dose of study therapy. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Limited extrahepatic disease would be allowed initially, that can be treated with stereotactic body radiation therapy (SBRT) or surgical resection prior to the start of tebentafusp. This concept is similar to the FOCUS trial - definition of "treatable" limited disease at the discretion of the PI.
* Ability to provide and understand written informed consent prior to any study procedures.

Exclusion Criteria:

* Life expectancy of less than 6 months.
* More than 50% of the liver volume replaced by tumor as measured by MRI.
* Extrahepatic disease as measured by CT of thorax abdomen and pelvis. (See inclusion criteria #10 above for limited treatable extrahepatic disease.)
* History of congestive heart failure, active cardiac conditions, including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), significant arrhythmias and severe valvular disease that precludes the use of general anesthesia.
* History or evidence of clinically significant pulmonary disease e.g. severe COPD that precludes the use of general anesthesia.
* Patients who are unable to undergo general anesthesia for any reason.
* Reduced renal function defined as Serum Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockcroft and Gault formula.
* Reduced hepatic function (defined as AST, ALT, bilirubin>2.5*ULN and PT-INR>1.5) or medical history of liver cirrhosis (Child-Pugh Class B or C) or evidence of portal hypertension by history, endoscopy or radiology.
* Hemoglobin <90 g/L or platelets <100x109/L or neutrophils <1.5x109/L.
* Use of live vaccines four weeks before the last study treatment.
* History of severe reactions to melphalan, heparin or iodine contrast. Iodine contrast reaction history patients permitted if patient will be treated with pre-meds, or if still problematic, treating physician may switch to MRI TAP.
* Known human immunodeficiency virus (HIV) infection, acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C.
* Active autoimmune disease or a documented history of autoimmune disease requiring active systemic immunosuppressive treatment. Type-1 diabetes, atopic dermatitis, and hypothyroidism are exceptions to this.
* A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Concomitant therapy with any other anti-cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications (other than physiologic (i.e., >10 mg) doses of steroids or as specified in exclusion #14) or use of other investigational drugs.
* Has a known additional malignancy that is progressing or requires active treatment.
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 150 days after the last dose of study drug.
* A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate in the opinion of the treating investigator.
* Previous treatment with PHP or tebentafusp.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 24 months
  PFS will be studied as time-to-event defined by the first documented disease progression or death due to any cause, whichever occurs first, from the start date of the study treatment. PFS will be determined based on tumor assessment (RECIST version 1.1 criteria).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 24 months
  ORR defined as the percentage of patients achieving a confirmed complete or partial response, as defined by RECIST version 1.1 criteria.
Clinical Benefit Rate (CBR) | Up to 24 months
  CBR defined as the percentage of patients achieving confirmed SD at 26 weeks, OR any confirmed CR or PR. As defined by RECIST version 1.1 criteria.
Hepatic PFS (hPFS) | Up to 24 months
  hPFS is defined as the time-to-event defined by the first documented disease progression in the liver or death due to any cause, whichever occurs first, from the start date of the study treatment. hPFS will be determined based on tumor assessment (RECIST version 1.1 criteria).
Overall Survival (OS) | Up to 24 months
  OS is calculated as the time-to-event defined by death due to any cause from the start date of the study treatment.
Melanoma-Specific Survival (MSS) | Up to 24 months
  MSS is calculated as the time-to-event defined by death due to uveal melanoma from the start date of the study treatment.
Time to Response (TTR) | Up to 24 months
  TTR calculated as the time-to-event defined by the first documented CR or PR from the start date of the study treatment.
Duration of Response (DOR) | Up to 24 months
  DOR calculated as the time-to-event defined by the first documented progression or death due to underlying cancer from the first document CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Zager, MD, FACS, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States